CLINICAL TRIAL: NCT02277886
Title: Clinical Trial: Esomeprazole Plus Alginate vs. Esomeprazole Alone for Treatment of Nighttime Reflux Symptom and GERD-related Sleep Disturbances in Patients With Erosive GERD
Brief Title: Esomeprazole Plus Alginate vs. Esomeprazole Alone for Treatment of Nighttime Reflux Symptom and Sleep Disturbances
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: TTY Biopharm (Industry)
Responsible Party: Principal Investigator, Cheng-Tang Chiu, Vice Director, Department of Internal Medicine, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALG-NR-14
Record Dates: First submitted 2014-10-02; First posted 2014-10-29 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Gastroesophageal Reflux Disease; Heartburn; Sleep Disturbance
Keywords: sodium alginate; esomeprazole; GERD
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn; Parasomnias | interventions — Alginates; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alginos plus Nexium (Experimental): sodium alginate 20ml (50mg/ml) once at bed time, and esomeprazole (40mg/tablet) 1 tablet once before breakfast, 4 weeks
  Interventions: Drug: sodium alginate; Drug: esomeprazole
- Nexium alone (Active Comparator): esomeprazole (40mg/tablet) 1 tablet once before breakfast, 4 weeks
  Interventions: Drug: esomeprazole

INTERVENTIONS:
Drug: sodium alginate — oral suspension, 50mg/ml, 20ml once at bed time
  Other Names: Alginos
  Arms: Alginos plus Nexium
Drug: esomeprazole — 40mg/tablet, one tablet once before breakfast
  Other Names: Nexium

SUMMARY:
Among those patients experienced GERD symptoms, up to 89% report nocturnal symptoms, resulting in poor sleep quality. Sodium alginate oral suspension (Alginos) is a medication indicated for the relief of gastroesophageal reflux symptoms. This multi-center, open-label, randomized trial intends to compare the addition of one dose Alginos (50mg/ml, 20ml) at bed time (Nexium plus Alginos), with no additional alginate treatment (Nexium alone), in erosive GERD patients taking Nexium (40mg/tablet) daily for 4 weeks. Efficacy endpoints include percentage of patients with relief or complete resolution of nighttime heartburn (or regurgitation), percentage of patients with relief or complete resolution of GERD-related sleep disturbance, the percentage of nights without nighttime heartburn (or regurgitation) over treatment period, change from baseline of the Pittsburgh Sleep Quality Index (PSQI) questionnaire total score, and change of the percentage of patients with relief of nighttime heartburn (or regurgitation) at post-treatment visit as compared to final visit in test group (Nexium plus Alginos). Safety endpoint is incidence of adverse events. The study hypothesis is that sodium alginate plus esomeprazole is superior to esomeprazole alone in relieving nighttime reflux symptoms and sleep disturbance in erosive GERD patients.

DETAILED DESCRIPTION:
This multi-center, open-label, randomized trial aims to compared the efficacy and safety profiles of sodium alginate oral suspension (50mg/ml) 20ml at bedtime with that of esomeprazole (40mg/tablet) 1 tablet once daily for the treatment of erosive GERD patients in Taiwan. Patients will be enrolled into study if they are diagnosed as GERD (grade A~D); with history of heartburn (or regurgitation) for ≥ 3 months before entering study; with history of GERD-related sleep disturbances for ≥ 1 month before entering study; with nighttime heartburn (or regurgitation) graded as moderate, or severe, on ≥ 3 nights in the last 7 days of screening period; with GERD-related sleep disturbances on ≥ 3 nights in the last 7 days of screening period; with the global PSQI score >5; and have signed the informed consent. Patients will be excluded if they are diagnosed as non-erosive GERD, Barrett's esophagus or esophageal stricture; with any conditions other than GERD that could be the primary cause of sleep disturbance; with active esophageal, gastric or duodenal ulcers; with history of esophageal, gastric or duodenal surgery; with active cancers of any kind; female patients who are pregnant or lactating; who were allergy to any of the study drugs; taking a proton pump inhibitor (PPI) within 7 days, or any prokinetic agent, H2-blocker, alginate preparations or antacid within 2 days before screening; with a history of drug addiction or alcohol abuse within the past 12 months; or with any other conditions or diseases that investigator considers it is not appropriate to enter the study. The primary efficacy endpoint is the percentage of patients with relief of nighttime heartburn (or acid regurgitation). The secondary efficacy endpoints are percentage of patients with complete resolution of nighttime heartburn (or regurgitation); percentage of patients with relief of GERD-related sleep disturbance; percentage of patients with complete resolution of GERD-related sleep disturbance; percentage of nights without nighttime heartburn (or regurgitation) over treatment period; change from baseline of the Pittsburgh Sleep Quality Index questionnaire total score (global PSQI score) at the end of study; and change of the percentage of patients with relief of nighttime heartburn (or acid regurgitation) at post-treatment visit (V4) as compared to final visit (V3) in test group (Nexium plus Alginos). The safety endpoint is incidence of adverse events. This study aims to prove that sodium alginate plus esomeprazole is superior to esomeprazole alone in relieving nighttime reflux symptoms and sleep disturbance in erosive GERD patients.

ELIGIBILITY:
Inclusion Criteria:

* Out -patients with age of 20-80 years old (inclusive) in Taiwan of both genders
* Patients who had been previously diagnosed as erosive GERD (i.e. grade A~D according to the modified Los-Angeles Classification. Endoscopic examination results within 21 days before randomization visit (V2) are acceptable.
* Patients with history of heartburn (or regurgitation) for ≥ 3 months before entering study
* Patients with history of GERD-related sleep disturbances for ≥ 1 month before entering study
* Patients with nighttime heartburn (or regurgitation) graded as moderate, or severe, on ≥ 3 nights in the last 7 days of screening period
* Patients with GERD-related sleep disturbances on ≥ 3 nights in the last 7 days of screening period
* Patients with the global PSQI score >5
* Patients have signed the informed consent form

Exclusion Criteria:

* Patients with non-erosive GERD, Barrett's esophagus or esophageal stricture
* Patients with any conditions other than GERD that could be the primary cause of sleep disturbance (e.g. sleep apnoea, obstructed airway, severe depression, severe anxiety, panic attacks, chronic obstructive pulmonary disease requiring oxygen therapy)
* Patients with active esophageal, gastric or duodenal ulcers
* Patients with history of esophageal, gastric or duodenal surgery
* Patients with active cancers of any kind
* Female patients who are pregnant or lactating
* Patients who were allergy to any of the study drugs
* Patients taken a proton pump inhibitor (PPI) within 7 days, or any prokinetic agent, H2-blocker, alginate preparations or antacid within 2 days before screening
* Patients with a history of drug addiction or alcohol abuse within the past 12 months
* Patients with any other conditions or diseases that investigator considers it is not appropriate to enter the study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with relief of nighttime heartburn (or acid regurgitation) | the last 7 days of study

SECONDARY OUTCOMES:
Percentage of patients with complete resolution of nighttime heartburn (or regurgitation) | the last 7 days of study
Percentage of Patients with relief of GERD-related sleep disturbance | the last 7 days of study
Percentage of Patients with complete resolution of GERD-related sleep disturbance | the last 7 days of study
The percentage of nights without nighttime heartburn (or regurgitation) over treatment period | the 28 days treatment period
Change from baseline of the Pittsburgh Sleep Quality Index questionnaire total score (global PSQI score) at the end of study | the 28 days treatment period
Change of the percentage of patients with relief of nighttime heartburn (or acid regurgitation) at post-treatment visit (V4) as compared to final visit (V3) in test group (Nexium plus Alginos) | 28 days after treatment stop

OTHER OUTCOMES:
Incidence of adverse events | the 28 days treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Tang Chiu, M.D., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taipei, Taiwan, Taiwan